CLINICAL TRIAL: NCT07037511
Title: Physiological, Sensory and Ergogenic Effects of Salbutamol - Implications for Athletic Screening and β2 Agonist Use in Sport
Brief Title: Effects of Salbutamol in Athletes and Implications for Screening and Sports
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jordan Guenette, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H24-01838
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Asthma; Healthy; Effect of Drug
Keywords: Exercise Physiology; Expiratory Flow Limitation; Non-Asthmatics; Beta2-Agonists
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salbutamol inhaler (Active Comparator): Participants will take four inhalations of salbutamol, with 60 seconds between each inhalation, totaling a therapeutic dose of 400µg of salbutamol prior to performing an incremental cardiopulmonary exercise test.
  Interventions: Drug: Salbutamol
- Placebo inhaler (Placebo Comparator): Participants will take four inhalations of placebo, with 60 seconds between each inhalation, prior to performing an incremental cardiopulmonary exercise test.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol — Meter-dose inhaler of salbutamol performed using large-volume spacer
  Arms: Salbutamol inhaler
Drug: Placebo — Meter-dose inhaler of placebo performed using large-volume spacer
  Arms: Placebo inhaler

SUMMARY:
β2-Agonists, commonly used to treat asthma, have also been used by athletes to enhance performance, leading to their ban by the International Olympic Committee in 1972. Research has shown non-asthmatics receive no benefit from these drugs at therapeutic dosages; however, many elite athletes still use them, and asthmatic athletes often win more Olympic medals. In some non-asthmatics, β2-agonists may improve breathing limitations during high intensity exercise, which may improve performance. Therefore, we aim to examine if there is a select group of non-asthmatic individuals who experience breathing limitations that may receive benefit from β2-agonists.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to examine the effects of β2-agonists on exercise performance in non-asthmatic male and female endurance athletes.

Hypothesis:

Our primary hypothesis is that ß2-agonists will improve exercise duration to a greater degree in athletes who experience expiratory flow limitation (EFL) compared to those who do not experience EFL. Additionally, female athletes will, on average, experience greater benefits with ß2-agonists due to a greater prevalence of EFL than males.

Justification:

While β2-agonists have historically been used by athletes as an ergogenic aid, systematic reviews indicate their ineffectiveness in improving aerobic performance. Consequently, the World Anti-Doping Agency (WADA) revised regulations to allow controlled use of specific β2-agonists. Despite a lack of evidence supporting their ergogenic benefits, positive tests for supratherapeutic doses of salbutamol among elite athletes, such as cyclist Chris Froome and cross-country skier Martin Johnsrud Sundby, suggests a belief in their performance-enhancing capabilities. Additionally, there is a physiological rationale for some non-asthmatics to benefit from these drugs. For instance, therapeutic doses of β2-agonists can induce bronchodilation, resulting in a ~5% increase in forced expiratory volume in one second (FEV1) in non-asthmatics. While this level of bronchodilation does not meet the diagnostic threshold for asthma, it holds potential for enhancing ventilatory responses in certain athletes. For example, a subset of non-asthmatic athletes who develop EFL during exercise, characterized by the inability to increase expiratory flows despite increases in expiratory effort, may derive greater benefits if the bronchodilation is sufficient to attenuate EFL. Indeed, experimental reduction of EFL via breathing a helium-oxygen gas mixture improves ventilatory responses, gas exchange, and endurance performance in non-asthmatics. We speculate that non-asthmatics experiencing EFL during exercise are likely to benefit more from β2-agonists than those who do not develop EFL.

Statistical Analysis:

The effects of salbutamol vs. placebo on exercise duration in all participants will be compared using a paired t-test. In all cases, a P-value < 0.05 will be considered statistically significant. A total of 64 participants (32 males and 32 females) will be recruited to adequately assess the effects of salbutamol on exercise tolerance, dyspnea, and related physiological variables.

ELIGIBILITY:
Inclusion Criteria:

* Aerobic capacity (V̇O2max) greater than 120% predicted
* Body mass index (BMI) > 18 and < 30 kg/m2
* Ability to read and understand English
* Currently training and/or competing in endurance sports (i.e. running or cycling)

Exclusion Criteria:

* Smoking history or currently smoking. Currently smoking is defined as regular use of cigarettes or cannabis at any point in the past year. History of smoking is defined as smoking more than 1 pack year for cigarettes or the equivalent in cannabis use measured as puffs per day / 200 (number of puffs in a pack of cigarettes).
* Use of cannabis within the past 30 days or has a smoking history of at least 1 pack year.
* Use of vaping devices or e-cigarettes in the past 30 days, or has used them more than 10 times in their lifetime.
* History or current symptoms of cardiopulmonary disease (excluding controlled asthma)
* Contraindications to exercise testing defined as anything that would prevent exercise under proper and safe conditions (e.g., a problem with the heart or lungs, muscle)
* Neuromuscular or musculoskeletal condition

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in time to exhaustion following salbutamol inhalation compared to placebo inhalation. | Up to 2 weeks
  Exercise duration will be measured during a time to exhaustion cardiopulmonary exercise test on a stationary cycle ergometer or treadmill.
Sex differences in time to exhaustion following salbutamol inhalation | Up to 2 weeks
  Exercise duration will be measured during a time to exhaustion cardiopulmonary exercise test on a stationary cycle ergometer or treadmill. Sexes will be compared within modality.

SECONDARY OUTCOMES:
To examine the effects of salbutamol on expiratory flow limitation in endurance athletes | Up to 2 weeks
  Expiratory flow limitation will be assessed by placing the tidal flow-volume loop within the maximal flow-volume loop during incremental cardiopulmonary exercise testing on a stationary cycle ergometer or treadmill.
To explore sex differences in dyspnea following salbutamol inhalation. | Up to 2 weeks
  Dyspnea will be assessed during and after both incremental and time to exhaustion cardiopulmonary exercise testing on a stationary cycle ergometer or treadmill with salbutamol.
To examine ventilatory responses of male and female endurance athletes to exercise with salbutamol. | Up to 2 weeks
  Ventilatory responses will be measured continuously throughout both incremental and time to exhaustion cardiopulmonary exercise testing on a stationary cycle ergometer or treadmill using a metabolic cart.
To explore the effects of salbutamol on exercise duration and expiratory flow limitation in both asthmatic and non-asthmatic individuals. | Up to 2 weeks
  A Eucapnic Voluntary Hyperpnea (EVH) test will be performed to assess airway hyperresponsiveness and classify participants as EVH-positive or EVH-negative. All participants will undergo the same cardiopulmonary exercise testing on a stationary cycle ergometer or a treadmill with salbutamol.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan A Guenette, PhD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada